CLINICAL TRIAL: NCT06458946
Title: Study the Postprandial Blood Glucose and Insulin in Different Fruit Snacks
Brief Title: Monitoring Postprandial Blood Glucose and Insulin in Fruit Snacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ocean Spray Cranberries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO-2405
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Blood Glucose; Blood Insulin
Keywords: blood glucose; metabolic health; cranberry fruit snacks

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Tested fruit bites are masked. Confection control is hard to mask (open label).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- First product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 5 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Fruit snack 1; Dietary Supplement: Fruit snack 2; Dietary Supplement: Fruit snack 3; Dietary Supplement: Fruit snack 4; Dietary Supplement: Fruit snack 5; Dietary Supplement: Confection control
- Second product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 5 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Fruit snack 1; Dietary Supplement: Fruit snack 2; Dietary Supplement: Fruit snack 3; Dietary Supplement: Fruit snack 4; Dietary Supplement: Fruit snack 5; Dietary Supplement: Confection control
- Third product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 5 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Fruit snack 1; Dietary Supplement: Fruit snack 2; Dietary Supplement: Fruit snack 3; Dietary Supplement: Fruit snack 4; Dietary Supplement: Fruit snack 5; Dietary Supplement: Confection control
- Fourth product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 5 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Fruit snack 1; Dietary Supplement: Fruit snack 2; Dietary Supplement: Fruit snack 3; Dietary Supplement: Fruit snack 4; Dietary Supplement: Fruit snack 5; Dietary Supplement: Confection control
- Fifth product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 5 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Fruit snack 1; Dietary Supplement: Fruit snack 2; Dietary Supplement: Fruit snack 3; Dietary Supplement: Fruit snack 4; Dietary Supplement: Fruit snack 5; Dietary Supplement: Confection control
- Sixth product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 5 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Fruit snack 1; Dietary Supplement: Fruit snack 2; Dietary Supplement: Fruit snack 3; Dietary Supplement: Fruit snack 4; Dietary Supplement: Fruit snack 5; Dietary Supplement: Confection control

INTERVENTIONS:
Dietary Supplement: Fruit snack 1 — Fruit snack with original level of sugar
Dietary Supplement: Fruit snack 2 — Fruit snack with reduced level of sugar
Dietary Supplement: Fruit snack 3 — Fruit snack with 0 added sugar - formulation 1
Dietary Supplement: Fruit snack 4 — Fruit snack with 0 added sugar - formulation 2
Dietary Supplement: Fruit snack 5 — Fruit snack from raisins
Dietary Supplement: Confection control — confection

SUMMARY:
The goal of this clinical trial is to compare the postprandial glucose and insulin responses after different fruit snacks compared to confection control in a healthy population

DETAILED DESCRIPTION:
Fruit snacks made form sweetened dried fruits are great sources of polyphenols, fiber, and other nutrients. The addition of sugar could help the taste, texture, and shelf life of this type of product. Fruit snacks with different levels of sugar were developed to meet various consumer needs and the postprandial glucose response in healthy population compared with confection control is of interest to study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 to ≤45 years of age at visit 1.
2. BMI ≥18.5 and <30.0 kg/m2 at visit 1.
3. Fasting capillary glucose <110 mg/dL at visit 1.
4. Willing to avoid consuming high-polyphenol containing foods for 48 h prior to each test visit.
5. Willing to abstain from alcohol consumption for 24 hours prior to each study visit.
6. Non-user of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months of visit 1, with no plans to begin use during the study period.
7. Willing to maintain habitual physical activity level throughout the duration of the study.
8. Willing to maintain habitual dietary pattern throughout the duration of the study, including stable intake of current vitamins, minerals, supplements and medications not interfering with study outcomes.
9. Score of 7 to 10 on the Vein Access Scale at visit 1.
10. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history.
11. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. History or presence of clinically important cardiac, renal, hepatic, endocrine, pulmonary, biliary, pancreatic, or neurological disorders that may affect the participant's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Investigator.
2. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at visit 1
3. Unstable use (initiation or change in dose) within 30 days of visit 1 of antihypertensive medications.
4. Unstable use (initiation or change in dose) within 30 days of visit 1 of thyroid hormone replacement medications.
5. Use of medications or supplements that may influence carbohydrate metabolism within 30 days of visit 1.
6. Extreme dietary habits (e.g., ketogenic, very high protein, very high fiber, vegan, vegetarian) at the discretion of the Clinical Investigator.
7. Weight loss or gain >4.5 kg in the 2 months prior to visit 1.
8. Currently, or planning to be, on a weight loss regimen during the study.
9. Use of weight loss medication within 90 d of visit 1.
10. History of gastrointestinal surgery for weight reducing purposes.
11. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
12. Known allergy or sensitivity to any ingredients or potential allergens contained in the study product.
13. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
14. History of any major trauma or major surgical event within 2 months of visit 1.
15. Blood donation >450 mL within 8 weeks of visit 2 or plans to donate blood or plasma during the study period.
16. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential with unstable use (initiation or change in dose) within 30 days of visit 1) of sex hormones for contraception.
17. Recent history of (within 12 months of screening; visit 1) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
18. Exposed to any non-registered drug product within 30 days prior to visit 1.
19. Any condition the Investigator believes would interfere with the participant's ability to provide informed consent or comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose iAUC - 2 hours | 2 hours
  The primary outcome variable will be glucose incremental area under the curve (iAUC) from pre-product consumption to 120 min (iAUC0-120 min)

SECONDARY OUTCOMES:
Blood glucose change | 2 hours
  Plasma glucose concentration change (Cmax - Cbaseline)
blood glucose time to max concentration | 2 hours
  Plasma glucose time to Cmax (Tmax)
Blood insulin | 2 hours
  Serum insulin iAUC, concentration change, time to the max concentration in 2 hours after consumption

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Shan, MD, Principal Investigator — Biofortis Innovation Services
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No